CLINICAL TRIAL: NCT03122366
Title: TLR4 Polymorphisms and Predisposition for Skin Cancer Development
Brief Title: TLR4 Polymorphisms and Risk of Skin Cancer
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Nabiha Yusuf, Associate Professor, University of Alabama at Birmingham
Other Study IDs: F080815001
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Skin Cancer
Keywords: single nucleotide polymorphisms; Toll-like receptor-4
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Detection of single nucleotide polymorphisms (SNP) — Asp299Gly SNP in the third exon of the TLR4 gene will be detected in blood

SUMMARY:
Toll-like receptors (TLRs) play a key role in the innate immune system. Toll-like receptor-4 (TLR4) in particular, appears to play a role in susceptibility to cancer. Of 44 identified SNPs (small nucleotide polymorphisms) in TLR4, the most common is an A-G substitution at nucleotide position +896, downstream of the cDNA start codon, a missense mutation which leads to an amino acid substitution Asp299Gly in the third exon of the TLR4 gene. Pre-clinical studies from our laboratory have shown an association of TLR4 with ultraviolet radiation induced skin cancer. Hence, in this study we will assess the pattern of TLR4 polymorphisms and susceptibility to skin cancer.

DETAILED DESCRIPTION:
Toll-like receptors (TLRs) play a key role in the innate immune system. Toll-like receptors generally, and TLR4 in particular, appear to play a role in cancer susceptibility as well as tumor immunosuppression and stromal invasion. Of 44 identified SNPs (small nucleotide polymorphisms) in TLR4, the most common is an A-G substitution at nucleotide position +896, downstream of the cDNA start codon, a missense mutation which leads to an amino acid substitution Asp299Gly in the third exon of the TLR4 gene, and which was later shown to co-segregate with SNP Thr399Ile-also in the third exon of TLR4.1 This SNP, present in 10% of the general population, has been found associated with gastric cancer, prostate cancer, and nasopharyngeal cancer.2-4 Pre-clinical studies from our laboratory have shown an association of TLR4 with ultraviolet radiation induced skin cancer. Hence, in this study we will assess the pattern of TLR4 polymorphisms and susceptibility to skin cancer.

ELIGIBILITY:
Inclusion Criteria:

* Male or female over the age of 50
* Fitzpatrick skin type I-IV

Exclusion Criteria:

* Tumor types other than basal cell carcinoma, squamous cell carcinoma and melanoma
* Chronic immunosuppression due to transplant antirejection regimen or HIV/AIDS
* Nevoid basal cell carcinoma syndrome, Cowden's syndrome, xeroderma pigmentosum or other syndrome with skin-cancer predisposition
* Known exposure to arsenic or ionizing radiation

Ages: 50 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 400 patients age 50 and older (case group) will be enrolled at the time of presentation for skin cancer excision surgery. These patients will be stratified into melanoma and non-melanoma skin cancer subgroups, and the non-melanoma subgroup will be further divided into prior and no prior history of skin cancer. All groups will have blood drawn at the time of enrollment. 400 patients age 50 and older (control group) with no personal history of skin cancer will be enrolled at our clinical trials unit. These patients will be stratified into family history and no family history of skin cancer subgroups, and will have blood drawn at the time of enrollment.
Sampling Method: Probability Sample
Enrollment: 392 (Actual)
Dates: Start 2009-02-02 (Actual); Primary Completion 2011-09-27 (Actual); Study Completion 2011-09-27 (Actual)

PRIMARY OUTCOMES:
single nucleotide polymorphism | once during the course of study
  TLR4 SNP Asp299Gly

CONTACTS AND LOCATIONS:
Overall Officials: Nabiha Yusuf, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The Kirklin Clinic, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No